CLINICAL TRIAL: NCT05510349
Title: Prevention of Per-partum Fetal Hypoxia: Measure of Placental Elasticity and Viscosity During Labor
Acronym: ELASTOLab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/652
Record Dates: First submitted 2022-08-08; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2021-10

CONDITIONS: Placental Elastography; Fetal Monitoring
MeSH Terms: interventions — Viscosity

STUDY DESIGN:
Intervention Model Description: Sonographic measure of placental elasticity and viscosity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All the patients (Experimental): Sonographic measure of placental elasticity and viscosity
  Interventions: Other: Sonographic measure of placental elasticity and viscosity

INTERVENTIONS:
Other: Sonographic measure of placental elasticity and viscosity — Sonographic measure of placental elasticity and viscosity

SUMMARY:
Fetal heart rate (FHR) monitoring during labor aims to detect fetuses at risk of intrapartum hypoxia in order to accelerate their birth before the constitution of sequelae such as anoxic encephalopathy and cerebral palsy. But the positive predictive value of FHR monitoring is low, and many second-line tests have been proposed but none of them has been proven to be conclusive. Measure of placental elasticity and viscosity during labor could be a new second line test to complete the FHR monitoring. Several studies have shown that placental elasticity is increased in case of gestational diabetes, preeclampsia, or intrauterine growth restriction, but no study has focused on placental elasticity during labor. The investigators hypothesize that placental elasticity and viscosity could reflect the quality of maternal-fetal exchanges during labor, and could help to detect fetus at risk of intrapartum hypoxia.

The first aim of this study is to describe the values of placental elasticity and viscosity during different points in the labor: beginning of the labor, beginning of the active phase of the first stage of labor, and passive phase of the second stage of labor.

Secondary aims of this study are: to describe the values of placental elasticity and viscosity in case of oxytocin infusion, in case of abnormal FHR, and ex-vivo after placental expulsion.

This unicentric observational prospective study will include 150 patients with singleton pregnancy, without pathology, with spontaneous labor at term.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* spontaneous labor at term
* body mass index < 30 at the beginning of the pregnancy
* anterior, lateral or fundal placenta
* epidural analgesia at the beginning of the labor
* normal fetal heart rate at the beginning of the labor

Exclusion Criteria:

* gestational diabetes
* preeclampsia
* intrauterine growth restriction

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Placental elasticity in kilopascals (kPa) | Day 1
  beginning of the labor
Placental viscosity in Pascal.seconde (Pa.s) | Day 1
  beginning of the labor
Placental elasticity in kilopascals (kPa) | Day 1
  beginning of the active phase of the first stage of labor
Placental viscosity in Pascal.seconde (Pa.s) | Day 1
  beginning of the active phase of the first stage of labor
Placental elasticity in kilopascals (kPa) | Day 1
  passive phase of the second stage of labor
Placental viscosity in Pascal.seconde (Pa.s) | Day 1
  passive phase of the second stage of labor

SECONDARY OUTCOMES:
Placental elasticity in kilopascals (kPa) | Day 1
  in case of oxytocin infusion
Placental viscosity in Pascal.seconde (Pa.s) | Day 1
  in case of oxytocin infusion
Placental elasticity in kilopascals (kPa) | Day 1
  in case of abnormal FHR
Placental viscosity in Pascal.seconde (Pa.s) | Day 1
  in case of abnormal FHR
Placental elasticity in kilopascals (kPa) | Day 1
  ex-vivo after placental expulsion
Placental viscosity in Pascal.seconde (Pa.s) | Day 1
  ex-vivo after placental expulsion